CLINICAL TRIAL: NCT04038684
Title: Healthy Eating, Activity and Reduction of Teen Stress
Acronym: HEARTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: Case Western Reserve University (Other); The Miriam Hospital (Other); Brown University (Other); Rhode Island Hospital (Other); University of North Carolina, Chapel Hill (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Amy Sato, Associate Professor of Psychological Sciences, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-201
Record Dates: First submitted 2019-07-12; First posted 2019-07-31 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Overweight and Obesity; Overweight Adolescents; Emotional Stress; Stress, Psychological; Eating Behavior
Keywords: Emotional Eating; Low-income; Mindfulness; Adolescent; Obesity; Weight Management; Stress; Pediatric
MeSH Terms: conditions — Overweight; Obesity; Stress, Psychological; Feeding Behavior; Emotional Eating

STUDY DESIGN:
Intervention Model Description: During the open trial, all participants will receive Mindfulness-Based Behavioral Weight Control (MBWC). During the RCT, participants will be randomly assigned to either MBWC or Standard Behavioral Weight Control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Weight Control (Experimental): All participants will be randomly assigned to a 12-session group-based Mindfulness-Based Weight Control (MBWC) intervention or a Standard Behavioral Weight Control (SBWC) intervention. Participants assigned to the MBWC intervention will receive mindfulness curriculum informed by Mindfulness-Based Stress Reduction plus the standard behavioral weight control components. Group sessions will be approximately 60 minutes each week. Outside of group sessions, participants will be asked to engage in dietary self-monitoring (MBWC and SBWC groups) and practice mindfulness skills (MBWC only).
  Interventions: Behavioral: Mindfulness-Based Weight Control (MBWC)
- Standard Behavioral Weight Control (Active Comparator): All participants will be randomly assigned to a 12-week group-based Mindfulness-Based Behavioral Weight Control (MBWC) intervention or a Standard Behavioral Weight Control (SBWC) intervention. Participants assigned to the SBWC intervention will receive the SBWC without mindfulness components. Each of the 12 group sessions will be approximately 60 minutes. Outside of group sessions, participants will be asked to practice dietary self-monitoring at home during the week.
  Interventions: Behavioral: Standard Behavioral Weight Control (SBWC)

INTERVENTIONS:
Behavioral: Mindfulness-Based Weight Control (MBWC) — Mindfulness-Based Weight Control will be administered over 12 group-based sessions with weekly home practice (e.g., mindfulness exercises, dietary self-monitoring, physical activity). All components of this telehealth intervention will be delivered via HIPAA-compliant videoconferencing software. Sessions will include BWC and mindfulness components. BWC components include: 1) a dietary plan based on a balanced, caloric deficit diet; 2) increasing physical activity; 3) behavioral components (e.g., self-monitoring, goal setting); and 4) minimal parent involvement (i.e., 3 parent sessions). Participants will be taught core mindfulness exercises (e.g., breath-awareness, body scan, mindful eating) while focusing attention on the present moment and non-judgmentally acknowledging thoughts, emotions, or sensations. Participants will learn informal mindful strategies for daily living, which are designed to increase awareness of emotions and their relation to emotional eating.
  Arms: Mindfulness-Based Weight Control
Behavioral: Standard Behavioral Weight Control (SBWC) — Standard Behavioral Weight Control will be administered over 12 group-based sessions with weekly home activities (dietary self-monitoring, physical activity). All components of this telehealth intervention will be delivered via HIPAA-compliant videoconferencing software. Group sessions will include SBWC component, including: 1) a balanced, caloric deficit diet; 2) incrementally increasing physical activity; 3) behavioral components (e.g., self-monitoring, goal setting, motivation, problem-solving, etc.); and 4) minimal parent involvement (i.e., 3 parent sessions).
  Arms: Standard Behavioral Weight Control

SUMMARY:
The goal of this study is to develop and pilot test a telehealth behavioral weight control intervention for adolescents from a low-income background that combines facets of mindfulness training with behavioral weight control. We aim to examine biological (e.g., weight) and behavioral (e.g., emotional eating, mindfulness) changes as a result of a 12-session mindfulness-based weight control intervention compared to a 12-session standard behavioral weight control intervention.

DETAILED DESCRIPTION:
The overarching aim of this study is to pilot and refine a novel Mindfulness-Based Weight Control (MBWC) intervention to improve weight management outcomes among adolescents (ages 13-18) who are overweight or obese and from a low-income background. First, we will pilot (open-trial) the MBWC intervention, with a focus on decreasing emotional eating, in an adolescent population. Second, we will conduct a randomized controlled trial of the 12-week MBWC intervention vs. a 12-week standard behavioral weight control intervention among adolescents who are overweight or obese and compare outcomes of the MBWC and control interventions. All components of this telehealth intervention will be delivered via HIPAA-compliant videoconferencing software. We are interested in examining change in biological and behavioral variables (e.g., body mass index normed for age and biological sex; perceived stress; eating and activity patterns; psychological function related to weight management) post-intervention and at three-month follow-up. Treatment satisfaction/treatment acceptability will be evaluated at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 13-18 years old
2. BMI in the overweight or obese range (≥ 85th%ile for age and sex)
3. speak English

Exclusion Criteria:

1. use of medications that have recently resulted in a change in eating or weight
2. cognitive impairment/developmental delay such that study procedures would be inappropriate
3. major psychiatric disorder (e.g. clinically severe depression, psychosis, anorexia nervosa, bulimia nervosa)
4. current participation in a weight loss program
5. pregnant or breastfeeding
6. medical condition known to impact weight or that would otherwise prevent participation

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 139 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Adolescent Body Mass Index (BMI) | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Objectively measured BMI/BMI z-score/BMI percentile for age and sex;
Change in Adolescent Emotional Eating | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Emotional Eating Scale for Children (EES-C) total score, which is derived from an average of all 26 items (range = 0-4). Higher scores indicate higher levels of emotional eating.
Change in Adolescent Perceived Stress | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Perceived Stress Scale (PSS) total score, which is derived from summing responses to all 10 items (range = 0-4 per item; 0-40 total). Higher scores indicate higher levels of stress.
Change in Adolescent Stress | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Adolescent Stress Questionnaire (ASQ) total score, which is derived from summing responses to all 58 items (range = 1-5 per item; 58-290 total). Higher scores indicate higher levels of stress.
Change in Adolescent Chronic Stress | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Chronic Stress Questionnaire for Children and Adolescents (CSQ-CA) total score, which is derived from summing responses to all 17 items (range = 1-4 per item; 17-68 total). Higher scores indicate more stress during the past 3 months.
Intervention Acceptability and Feasibility | End of treatment (approx 14 weeks after baseline)
  Acceptability and feasibility of the mindfulness-based behavioral weight control intervention will be measured by session attendance, dietary self-monitoring logs, and attrition rates.

SECONDARY OUTCOMES:
Change in Adolescent Eating Pathology and Symptomology | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Youth Eating Disorder Examination-Questionnaire (YEDE-Q) global score, which is derived by averaging the 4 subscales of the YEDE-Q (Restraint, Eating Concern, Shape Concern, and Weight Concern). The range for the total score is 0 to 6, with higher scores indicating more severe eating pathology.
Change in Adolescent Eating Behaviors | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Three Factor Eating Questionnaire (TFEQ), which includes subscales representing uncontrolled eating, cognitive restraint, and emotional eating. Each of the 18 items are rated on a scale of 1-4. Higher scores indicate higher levels of each eating behavior.
Change in Adolescent Emotion Regulation | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) includes two subscales representing emotion regulation strategies (Suppression and Reappraisal). Responses to all 10 items (range = 1-7 per item) are summed to calculate each subscale. Higher scores indicate higher use of each emotion regulation strategy.
Change in Adolescent Mindfulness | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Child and Adolescent Mindfulness Measure (CAMM) total score, which is derived from reverse scoring and summing responses to all 25 items (range = 0-4 per item; 0-100 total). Higher scores indicate higher acceptance and mindfulness.
Change in Adolescent Mindful Attention Awareness | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Mindfulness Attention Awareness Scale - Adolescent (MAAS-A) total score, which is derived from summing responses to all 15 items (range = 1-6 per item; 15-90 total). Higher scores indicate higher trait mindfulness.
Change in Adolescent Quality of Life - Adolescent Report | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Sizing Me Up total score, which is derived from responses on 22 items (range = 1-4). Raw scores are converted to a scaled score from 0-100, with higher scores indicating greater quality of life.
Change in Adolescent Quality of Life - Parent/Caregiver Report | baseline to intervention completion (approx 14 weeks), baseline to 3-month follow-up (approx 26 weeks), and intervention completion to 3-month follow-up.
  Sizing Them Up total score, which is derived from responses on 28 items (range = 1-4). Raw scores are converted to a scaled score from 0-100, with higher scores indicating greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Amy F Sato, PhD, Principal Investigator — Kent State University
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No